CLINICAL TRIAL: NCT02728037
Title: Randomized Control Trial of Magnesium-Based Trigger Point Injections vs. Lidocaine-Only Trigger Point Injections for Relief of Chronic Myofascial Pelvic Pain
Brief Title: Magnesium-Based Trigger Point Injections for Relief of Chronic Myofascial Pelvic Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low Enrollment, Adoption of investigational treatment into standard practice at our center.
Sponsor: Queen's University (Other)
Collaborators: Hotel Dieu Hospital (Other)
Responsible Party: Principal Investigator, Jessica Pudwell, Research Assistant, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OBGY-276-15
Record Dates: First submitted 2015-10-26; First posted 2016-04-05 (Estimated); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Pelvic Pain
Keywords: Myofascial Trigger Points; Myofascial Pain; Intramuscular Anesthetic Injection
MeSH Terms: conditions — Pelvic Pain | interventions — Lidocaine; Magnesium Sulfate; Bicarbonates; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Magnesium-Based Injection Formulation (Experimental): Examination will involve systematic palpation of the 3 distinct levels of pelvic musculature. Injections into level 1 and level 2 muscles will be done under ultrasound guidance. Level 3 injections will be facilitated with a trumpet guide when needed. As the pelvic muscle trigger points are identified they will be injected with 2-3ml of the prepared injection formulation. The investigator will continue until no further trigger points can be identified, a maximum dose of lidocaine has been used, or the participant indicates they wish to stop. The maximum dose of lidocaine is 5mg per kg of body weight (280 mg of lidocaine in a 55kg woman or approximately 40cc of the final mixture).
  Interventions: Procedure: Magnesium-Based Injection Formulation; Drug: lidocaine; Drug: magnesium sulfate, bicarbonate, dextrose.
- Lidocaine-Only Injection Formulation (Active Comparator): Examination will involve systematic palpation of the 3 distinct levels of pelvic musculature. Injections into level 1 and level 2 muscles will be done under ultrasound guidance. Level 3 injections will be facilitated with a trumpet guide when needed. As the pelvic muscle trigger points are identified they will be injected with 2-3ml of the prepared injection formulation. The investigator will continue until no further trigger points can be identified, a maximum dose of lidocaine has been used, or the participant indicates they wish to stop. The maximum dose of lidocaine is 5mg per kg of body weight (280 mg of lidocaine in a 55kg woman or approximately 40cc of the final mixture).
  Interventions: Procedure: Lidocaine-Only Injection Formulation; Drug: lidocaine
- Wait-Listed Patients (No Intervention): This arm is a non-randomized, no-treatment arm consisting of women who are on the waiting list for the chronic pain clinic.

INTERVENTIONS:
Procedure: Magnesium-Based Injection Formulation — Each study kit will include 4 10cc syringes containing 7ml of 1% lidocaine, and 3 numbered glass vials. For those in the magnesium-based injection formulation arm the glass vials will be prepared as follows; 1) 10ml of 50% magnesium sulfate, 2) 20ml of 8.4% bicarbonate, and 3) 20ml of 50% dextrose.
  At the visit a study investigator will mix 2cc of vial 1, 5cc of vial 2 and 5cc of vial 3, for a total of 12cc of additive mixture. 3cc of this additive mixture will be then drawn in to each of the 4 pre-packaged lidocaine syringes, for a total of 10cc of final mixture per syringe. The concentration of components in the final mixture is 0.7% lidocaine, 0.8% sodium bicarbonate, 6.0% dextrose, and 2.5% magnesium sulfate.
  Arms: Magnesium-Based Injection Formulation
Procedure: Lidocaine-Only Injection Formulation — Each study kit will include 4 10cc syringes containing 7ml of 1% lidocaine, and 3 numbered glass vials. For those in the lidocaine-based injection formulation arm the glass vials will be prepared as follows; 1) 10ml of 0.9% sodium chloride, 2) 20ml of 0.9% sodium chloride, and 3) 20ml of 0.9% sodium chloride.
  At the visit a study investigator will mix 2cc of vial 1, 5cc of vial 2 and 5cc of vial 3, for a total of 12cc of additive mixture. 3cc of this additive mixture will be then drawn in to each of the 4 pre-packaged lidocaine syringes, for a total of 10cc of final mixture per syringe. The concentration of components in the final mixture is 0.7% lidocaine.
  Arms: Lidocaine-Only Injection Formulation
Drug: lidocaine
  Arms: Lidocaine-Only Injection Formulation; Magnesium-Based Injection Formulation
Drug: magnesium sulfate, bicarbonate, dextrose.
  Arms: Magnesium-Based Injection Formulation

SUMMARY:
This study will be a randomized, controlled, double-blinded, single-centre superiority trial with two parallel groups. The primary outcome will be average myofascial pelvic pain in the two weeks following final injection treatment as assessed using the visual analogue scale. Randomization will be performed as block randomization with a 1:1 allocation ratio, stratified based on opioid use at the time of study enrollment. In total, 60 participants will be recruited and randomized, with 30 being assigned to each treatment arm. The study will be restricted such that none of the participants enrolled will be current concomitant opioid users (for any reason) and will not have used opioid drugs within the 3 months preceding enrollment in the study.

A third non-randomized arm of 30 participants who are on the waiting list for the chronic pain clinic will be enrolled and compared to the two randomized arms. Among this patient population and in the setting of the Chronic Pain Clinic it was determined that it would not be acceptable to randomize participants to a no-treatment control group. As such, an active treatment is being used as comparator in the randomized trial. In order to assess participants in the absence of treatment this third non-randomized arm will serve as a no-treatment control group.

Eligibility criteria for this third arm is the same as the main study, except for the restriction by opioid use status. Participation in this third arm will not exclude a participant from randomization into one of the two main arms of the study. Therefore, across the three arms, up to 90 patients will be enrolled in this study.

DETAILED DESCRIPTION:
Study Setting: This study will be conducted at the Chronic Pain Clinic at Hotel Dieu Hospital and the General Gynecology Clinic at Kingston General Hospital in Kingston, Ontario, Canada. All of the physicians who provide trigger point injection treatment for chronic pelvic pain in the Chronic Pain Clinic have agreed to participate as co-investigators in this study (RN, RH, and SC). Women are referred to this clinic for treatment of chronic pelvic pain by both primary care providers and gynecologists in the Kingston and surrounding area. Two of the investigators (RN and SC) see patients in the General Gynecology Clinic for assessment and management of chronic pelvic pain. Both investigators regularly refer patients to the Chronic Pain Clinic for consideration of trigger point injections.

Participant Timeline: Participants in this study will be followed for a total of 8 treatments and 9 study visits over a period of 12 weeks. Participants in the third wait-listed arm of the study will be followed for 3 visits over a period of 12 weeks.

Treatment Arms, Baseline Visit & Treatment 1: At the baseline study visit a research nurse will administer a questionnaire in order to obtain a thorough medical history and collect information on participant demographics. The research nurse will then administer the VAS pain scale and pelvic pain specific functional questionnaire based on the participant's experiences in the week preceding the baseline visit and the WHOQOL-BREF based on the participant's experiences in the 4 weeks preceding the baseline visit. A study investigator will then mix and administer the trigger point injections. The research nurse will remain present for the treatment to assist with recording and administer the VAS pain scale for procedural discomfort immediately following completion of treatment.

Treatment Arms, Follow Up Visits & Treatments 2-8: In total, participants will be seen for 7 follow up visits with additional treatment. Visits 2 through 4 will be done on a weekly basis and visits 5 through 8 will be done bi-weekly, for a total time of 11 weeks. At these visits a research nurse will administer the VAS pain scale and pelvic pain specific functional questionnaire based on the participant's experiences in the week preceding the visit. The research nurse will ask further questions about concomitant medication usage and screen participants for any adverse event or injection-associated complications. In addition at visit 5 the research nurse will administer the WHOQOL-BREF. A study investigator will then mix and administer the trigger point injections. The research nurse will remain present for the treatment to assist with recording and administer the VAS pain scale for procedural discomfort immediately following completion of treatment.

Treatment Arms, Final Study Visit 9: For participants who undergo a full course of treatment the final study visit will be visit 9 and will occur 12 weeks after the baseline visit. If a woman chooses to conclude treatment early, for any reason, then the final visit will occur earlier than 12 weeks. However, the final visit must always be done at least 1 week after the final trigger point injection treatment. At the final study visit a research nurse will administer the VAS pain scale and pelvic pain specific functional questionnaire based on the participant's experiences in the week preceding the visit and the WHOQOL-BREF based on the participant's experiences in the 4 weeks preceding the visit. The research nurse will ask further questions about concomitant medication usage and screen participants for any adverse event or injection-associated complications. In order to assess blinding participants will be asked which treatment they believed they received and their reasons for this belief. Participants will also be asked if they would recommend the treatment to others experiencing myofascial pelvic pain. Finally, participants will be offered continuation of treatment under the care of the primary investigator with an injection formulation of their choosing if they are still experiencing myofascial pelvic pain.

Wait-List Arm, Baseline, Follow Up and Final Study Visit: At the baseline study visit a research nurse will administer a questionnaire in order to obtain a thorough medical history and collect information on participant demographics. The research nurse will then administer the VAS pain scale and pelvic pain specific functional questionnaire based on the participant's experiences in the week preceding the baseline visit and the WHOQOL-BREF based on the participant's experiences in the 4 weeks preceding the baseline visit. The research nurse will ask further questions about concomitant medication usage. A follow up visit will be completed 5 weeks after the baseline visit. At this visit a research nurse will administer the VAS pain scale and pelvic pain specific functional questionnaire based on the participant's experiences in the week preceding the visit and the WHOQOL-BREF based on the participant's experiences in the 4 weeks preceding the visit. The research nurse will ask further questions about concomitant medication usage. For participants who are on the wait-list for at least 12 weeks the final study visit will occur 12 weeks after the baseline visit. If a woman is on the wait-list for under 12 weeks then the final study visit will occur at her first visit to the Chronic Pain Clinic. At the final study visit a research nurse will administer the VAS pain scale and pelvic pain specific functional questionnaire based on the participant's experiences in the week preceding the visit and the WHOQOL-BREF based on the participant's experiences in the 4 weeks preceding the visit. The research nurse will ask further questions about concomitant medication usage.

ELIGIBILITY:
Potential participants will be screened for eligibility based on the following inclusion and exclusion criteria. All of the following criteria will be used to screen participants for enrollment and randomization into one of the two treatment arms. All of the following criteria except for inclusion criteria number 2 and exclusion criteria number 10 will be used to screen participants for enrollment into the third wait-listed patient arm. These eligibility exceptions are necessary for the third arm as opioid medication may be introduced as temporary medical management for the condition while patients wait for acceptance into the Chronic Pain Clinic.

Inclusion Criteria:

1. Patients with a clinical diagnosis of chronic pelvic pain lasting 6 months or greater
2. Not an opioid user: no opioid analgesic use for relief of chronic pelvic pain within the last 3 months

Exclusion Criteria:

1. Age <18 years or age >65 years at the time of study enrollment
2. Pregnancy (currently pregnant or planning to become pregnant during the study period)
3. Known allergy or sensitivity to local anesthetics, dextrose, sodium bicarbonate or magnesium-sulfate
4. A clinical diagnosis of fibromyalgia
5. Having received previous trigger point injections of any formulation for pelvic pain
6. Bleeding disorders (including, but not limited to, hemophilia and von Willebrand disease)
7. Currently receiving anticoagulation therapy (including, but not limited to, coumadins, heparin and its derivatives, direct thrombin inhibitors, and anti-thrombin protein therapeutics; use of low dose aspirin is permitted)
8. Living greater than 50 km to the pain clinic at Hotel Dieu Hospital in Kingston, Ontario, Canada
9. Current opioid analgesic use for a reason other than chronic pelvic pain (including, but not limited to, ongoing opioid dependency or relief of other pain symptoms)
10. Recent opioid analgesic use for relief of chronic pelvic pain; defined as use within the last 3 months but not within the last 2 weeks prior to enrollment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-04; Primary Completion 2020-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Mean Change in Average Pelvic Pain | 12 Weeks
  The primary outcome measure a comparison of the two treatment arms. It is the mean change in average pain in the week preceding the study visit, from baseline to final visit, as measured by the visual analogue pain scale. Using this scale participants rate their average pain over the last week on a scale from 0 to 10 by drawing an "x" on the horizontal line. This line is 10cm long and the participant's pain level is measured using a ruler to the millimeter mark and translated to a score out of 100mm. If the "x" falls between millimeter marks on the ruler the reader will round up to the nearest mark.

SECONDARY OUTCOMES:
Mean Change in Functional Pelvic Pain | 12 Weeks
  A comparison of the two treatment arms. Function will be scored at each visit using a validated functional pelvic pain scale. The functions of bladder, bowel, intercourse, walking, running, lifting, working and sleeping are each rated on a Likert scale from 0 to 4. With 0 corresponding to no pain and normal function and 4 corresponding to an inability to function because of pain. Participants are asked to rank these functions based on when their pain was at its worst in the last week. Both individual functions and overall function score will be considered.
Mean Change in Quality of Life | 12 Weeks
  A comparison of the two treatment arms. Quality of life will be scored using the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF) at the baseline, fifth, and final visit. The WHOQOL-BREF assesses quality of life in 4 domains of physical health, psychological health, social relationships, and environment through a series of 26 questions using a Likert scale from 1 to 5. Changes in each of these 4 domains over the course of treatment will be considered.
Change in Average Daily Concomitant Opioid Analgesic Usage | 12 Weeks
  At each study visit participants will be asked to report their average daily concomitant analgesic medication usage during the preceding week, which will be recorded in the concomitant medication log. Type of medication, dosage and frequency of usage will be recorded. This comparison will focus on opioid medication usage and the summary measure of number of days in the preceding week that at least one dose of an opioid medication was required will be used. If a participant required at least one dose of opioid medication every day of the preceding week then they will be assigned a summary measure of 7. If they only required at least one dose of opioid medication on two days in the preceding week then they will be assigned a summary measure of 2. Changes in these summary measures over the 12 week course of treatment will be compared between the two treatment arms.
Procedural Pain | 12 weeks
  A comparison of the two treatment arms. At each visit participants will be asked to report the level of pain experienced during administration of injections. Immediately following administration, participants will report this using the same visual analogue scale used to measure the primary outcome. Each participants average procedural pain score over the course of treatment will be calculated. These average procedural pain will be compared between treatment groups.
Time to Resolution of Symptoms | 12 Weeks
  A comparison of the two treatment arms. The time to resolution of symptoms to a manageable level in weeks of treatment will be compared between groups. Participants will stop receiving treatment either at their 8th visit (12 weeks from baseline) or earlier if they choose. Only those women who indicate that their pain has reached a manageable level at the time of treatment conclusion will be included in this analysis.
Complications and/or Adverse Events | 12 Weeks
  A comparison of the two treatment arms. At each study visit participants will be asked about any complications or adverse events that they may have experienced. Participants will also be monitored for complications and adverse events during the course of treatment at the pain clinic. The type and frequency of complications and adverse events will be compared between groups.
Comparison with the Wait-List Arm for the Primary Outcome: Mean Change in Average Pelvic Pain | 12 Weeks
  The primary outcome of mean change in average pain in the week preceding the study visit, from baseline to final visit, as measured by the visual analogue pain scale will be compared among the 3 study arms. The wait-listed arm will serve as a non-randomized, no-treatment comparison group.
  The primary outcome measure is the mean change in average pain in the week preceding the study visit, from baseline to final visit, as measured by the visual analogue pain scale. Using this scale participants rate their average pain over the last week on a scale from 0 to 10 by drawing an "x" on the horizontal line. This line is 10cm long and the participant's pain level is measured using a ruler to the millimeter mark and translated to a score out of 100mm. If the "x" falls between millimeter marks on the ruler the reader will round up to the nearest mark.
Comparison with the Wait-List Arm for the Secondary Outcome: Mean Change in Functional Pelvic Pain | 12 Weeks
  The wait-listed arm will serve as a non-randomized, no-treatment comparison group. A comparison of the 3 study arms will be completed.
  Function will be scored at each visit using a validated functional pelvic pain scale. The functions of bladder, bowel, intercourse, walking, running, lifting, working and sleeping are each rated on a Likert scale from 0 to 4. With 0 corresponding to no pain and normal function and 4 corresponding to an inability to function because of pain. Participants are asked to rank these functions based on when their pain was at its worst in the last week. Both individual functions and overall function score will be considered.
Comparison with the Wait-List Arm for the Secondary Outcome: Mean Change in Quality of Life | 12 Weeks
  The wait-listed arm will serve as a non-randomized, no-treatment comparison group. A comparison of the 3 study arms will be completed.
  A comparison of the two treatment arms. Quality of life will be scored using the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF) at the baseline, fifth, and final visit. The WHOQOL-BREF assesses quality of life in 4 domains of physical health, psychological health, social relationships, and environment through a series of 26 questions using a Likert scale from 1 to 5. Changes in each of these 4 domains over the course of treatment will be considered.
Comparison with the Wait-List Arm for the Secondary Outcome: Change in Average Daily Concomitant Opioid Analgesic Usage | 12 Weeks
  The wait-listed arm will serve as a non-randomized, no-treatment comparison group. A comparison of the 3 study arms will be completed.
  At each study visit participants will be asked to report their average daily concomitant analgesic medication usage during the preceding week, which will be recorded in the concomitant medication log. Type of medication, dosage and frequency of usage will be recorded. This comparison will focus on opioid medication usage and the summary measure of number of days in the preceding week that at least one dose of an opioid medication was required will be used. Changes in these summary measures over the 12 week course of treatment will be compared between the two treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Romy Nitsch, MD, MHSc, Principal Investigator — Queen's University
Locations (1):
- Department of Obstetrics & Gynecology, Queen's Unviersity, Kingston, Ontario, Canada

REFERENCES:
- [Background] Jarrell JF, Vilos GA. Consensus Guidelines for the Management of Chronic Pelvic Pain: SOGC Clinical Practice Guidelines. No 164, Part 1 of 2, August 2005.
- [Derived] Leitch J, Webb A, Pudwell J, Chamberlain S, Henry R, Nitsch R. Magnesium-Based Trigger Point Infiltrations Versus Local Anaesthetic Infiltrations in Chronic Pelvic Myofascial Pain: A Randomized, Double-Blind, Controlled Study. J Obstet Gynaecol Can. 2022 Aug;44(8):877-885. doi: 10.1016/j.jogc.2022.02.129. Epub 2022 Mar 24. PMID 35339694